CLINICAL TRIAL: NCT05894642
Title: Determination and Characterization of Persistent Musculoskeletal Pain in Covid-19 Patients in Primary Care.
Brief Title: Characterization of Long Covid Pain in Primary Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Laura Barrero Santiago, Phd Candidate, University of Valladolid
Other Study IDs: LGCOVIDCS
Record Dates: First submitted 2023-06-06; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Long COVID; Chronic Pain; Musculoskeletal Pain
Keywords: Long COVID; Chronic Pain; Musculoskeletal pain; Primary health care; Psychological factors
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- Long Covid Pain Patients
  Interventions: Behavioral: 0
- Control Group, healthy people: Patients that had had Covid-19 but did not developed chronic pain or other chronic symptoms.

INTERVENTIONS:
Behavioral: 0 — It is a case-control study, cross-sectional, so there is no intervention possible.
  Groups: Long Covid Pain Patients

SUMMARY:
Justification: among the sequelae of Covid-19 in clinical practice we frequently find persistent neuromusculoskeletal pain. Prevalence data and the underlying mechanisms of such pain are very limited in the scientific literature. Therefore, with this research we will try to answer these questions.

Main objective: to determine and characterize persistent musculoskeletal pain in Covid-19 patients.

Method: two phases. First, a descriptive cross-sectional study will be carried out to estimate the prevalence of Long Covid Pain (LCP). Second phase, a case-control study will be carried out using the sample obtained in the first phase as the population. The sample will be divided into two groups: post-Covid-19 patients with LCP and post-Covid-19 patients without persistent pain (control group). The two groups will be matched according to sex, age and level of severity of the pathology.

An assessment and comparison between groups will be made of the following variables: central sensitization, healthy physical condition and blood test values, which will be evaluated by means of physical examination, questionnaires and laboratory tests.

Applicability of the results: this is a pioneering project at the national level, which would determine more reliably the prevalence of LCP in postcovid and could be a first step in the search for the best therapeutic strategies for these patients. This would help to improve the quality of life of these patients and to better manage the social and healthcare resources used in their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had Covid-19, with a confirmatory PCR+ test or positive antigen test and recorded in their primary care medical record.
* Subjects between 18-70 years old.
* Musculoskeletal pain of more than 12 weeks of evolution since the beginning of the infection.
* Agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* History of chronic musculoskeletal pain of more than 12 weeks of evolution prior to Covid-19.
* History of diagnosed major depression.
* Having a diagnosis of fibromyalgia prior to Covid-19 infection.
* Pregnancy.
* Pain of oncologic origin.
* Fracture or surgical intervention on the spine in the last year.
* Bladder or bowel incontinence.
* Saddle anesthesia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Long Covid Pain Patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QoL) | 1 day
  EQ-5D questionnaire (Qualitave of Life 5 Dimension): The EQ-5D-3L is a brief multi-attribute health status measure composed of five questions with Likert response options (descriptive system) and a visual analogue scale (EQ-VAS). The descriptive system covers five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with three levels of severity in each dimension (no problems, some problems, and extreme problems).

SECONDARY OUTCOMES:
Pain Intensity | 1 day
  Visual Analog Scale, VAS (0-100mm).
Areas of pain | 1 day
  body chart, McGill questionnaire
Quantitative sensory tests | 1 day
  temporal summation, pain detection to pressure and conditioned modulation test
Handgrip Strength assessment | 1 day
  With a manual dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Valladolid, Valladolid, Spain